CLINICAL TRIAL: NCT05491876
Title: Comparison Of Active Cycle Of Breathing Technique And Breathing Exercises On Oxygen Saturation And Pulmonary Function Test In Post ICU COVID-19 Patients
Brief Title: Active Cycle Of Breathing Technique Verses Breathing Exercises In Post ICU COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0333
Record Dates: First submitted 2022-07-24; First posted 2022-08-08 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Post Covid-19 Patients
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: The study came to the conclusion that both techniques, breathing exercises with and without ACBT were beneficial in raising PaO2, FEV1, FVC, and the FEV1/FVC ratio as well as oxygen saturation.
  However, based on their mean differences, ACBT with breathing exercises was more beneficial in terms of the indicated end measures.
Who Masked: Participant
Masking Description: This evidence supports current study that the use of ACBT exercises with Breathing exercises is helpful to improve respiratory performance.
  single blinded study only participant blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest physiotherapy with breathing exercises and ACBT (Experimental): Group A will recieve chest physiotherapy with breathing exercises and ACBT.
  Interventions: Other: Chest physiotherapy with breathing exercises and ACBT
- Chest physiotherapy with breathing exercises (Experimental): Group B will receive chest physiotherapy with breathing exercises.
  Interventions: Other: Chest physiotherapy with breathing exercises

INTERVENTIONS:
Other: Chest physiotherapy with breathing exercises and ACBT — Group A got chest physiotherapy with breathing exercises and ACBT
  Other Names: ACTIVE CYCLE OF BREATHING TECHNIQUE (ACBT)
  Arms: Chest physiotherapy with breathing exercises and ACBT
Other: Chest physiotherapy with breathing exercises — Group B got chest physiotherapy with breathing exercises.
  Arms: Chest physiotherapy with breathing exercises

SUMMARY:
The experiment was randomized and controlled. To create groups A and B,48 individuals were selected by sample selection criteria. Evaluation of oxygen saturation and pulmonary function tests were taken using a pulse oximeter and spirometer. Group A got chest physiotherapy with breathing exercises and ACBT whereas Group B got chest physiotherapy with breathing exercises. The treatment took 15-30 minutes and consisted of one session per day, treatment was given 6 days a week for up to 2 weeks and examined by using SPSS 22.

DETAILED DESCRIPTION:
The experiment was randomized and controlled. To create groups A and B,48 individuals were selected by sample selection criteria. Evaluation of oxygen saturation and pulmonary function tests were taken using a pulse oximeter and spirometer. Group A got chest physiotherapy with breathing exercises and ACBT whereas Group B got chest physiotherapy with breathing exercises. The treatment took 15-30 minutes and consisted of one session per day, treatment was given 6 days a week for up to 2 weeks and examined by using SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* Adult population

  * Age limit 18 -50
  * All patients positive with confirmed COVID-19 by polymerase chain reaction (PCR) test and chest computed tomography scan (CT-scan)

Exclusion Criteria:

* The patient cannot take part in the trial if they have any kind of muscular-skeletal issue.

  * COVID-19-related intubation history
  * A clear clinical mental or cognitive disability of any kind.
  * Patient on ventilator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
SPIROMETRY | 4 weeks
  Spirometry is a simple test used to help diagnose and monitor certain lung conditions by measuring how much air you can breathe out in one forced breath. In a spirometry test, while you are sitting, you breathe into a mouthpiece that is connected to an instrument called a spirometer. The spirometer records the amount and the rate of air that you breathe in and out over a period of time. When standing, some numbers might be slightly different.
PULSE OXIMETRY | 4 weeks
  pulse oximetry is a painless, noninvasive method of measuring the saturation of oxygen in a person's blood. Oxygen saturation is a crucial measure of how well the lungs are working. When we breathe in air, our lungs transmit oxygen into tiny blood vessels called capillaries. A normal pulse oximeter reading for your oxygen saturation level is between 95% and 100%. If you have a lung disease such as COPD or pneumonia, your normal oxygen saturation level may be lower.

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, MS.CPPT, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gastaldi AC, Paredi P, Talwar A, Meah S, Barnes PJ, Usmani OS. Oscillating Positive Expiratory Pressure on Respiratory Resistance in Chronic Obstructive Pulmonary Disease With a Small Amount of Secretion: A Randomized Clinical Trial. Medicine (Baltimore). 2015 Oct;94(42):e1845. doi: 10.1097/MD.0000000000001845. PMID 26496331
- [Background] van Mourik Y, Rutten FH, Bertens LCM, Cramer MJM, Lammers JJ, Gohar A, Reitsma JB, Moons KGM, Hoes AW. Clinical research study implementation of case-finding strategies for heart failure and chronic obstructive pulmonary disease in the elderly with reduced exercise tolerance or dyspnea: A cluster randomized trial. Am Heart J. 2020 Feb;220:73-81. doi: 10.1016/j.ahj.2019.08.021. Epub 2019 Sep 1. PMID 31790904
- [Background] Gephine S, Mucci P, Grosbois JM, Maltais F, Saey D. Physical Frailty in COPD Patients with Chronic Respiratory Failure. Int J Chron Obstruct Pulmon Dis. 2021 May 17;16:1381-1392. doi: 10.2147/COPD.S295885. eCollection 2021. PMID 34045852